CLINICAL TRIAL: NCT03935503
Title: COMPARISON OF LAPAROSCOPIC TOTAL EXTRAPERITONEAL HERNIA REPAIR AND LICHTENSTEIN HERNIA REPAIR FOR SEXUAL, SENSORY, LIFE QUALITY AND URINARY FUNCTIONS
Brief Title: COMPARISON OF LAPAROSCOPIC TOTAL EXTRAPERITONEAL HERNIA REPAIR AND LICHTENSTEIN HERNIA REPAIR
Acronym: HERNIA
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ANIL ERGIN, Dr Anil ERGIN , General Surgery , Asistant doctor, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: ANIL ERGIN1
Record Dates: First submitted 2019-04-21; First posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-05

CONDITIONS: Inguinal Hernia
Keywords: Quality of life; Inguinal Hernia; Lichtenstein repair; Sexual Function; Total Extraperitoneal Repair
MeSH Terms: conditions — Hernia, Inguinal | interventions — tetraethylpyrazine

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Total Extraperitoneal Repair: Laparoscopic Total Extraperitoneal (TEP) method was performed to repair inguinal hernia . Patients were evaluated preoperatively, at 1 month and 6 months postoperatively, International Sexual Function Index (IFIF), International Prostatic Symptom Score, SF-36 Quality of Life Scale, Visual Analog Pain Scale, Beck Depression Scale, Inguinal Region Discrimination Test ( DT), DN4 Neuropathic Pain Survey, Uroflowmetry and FSH, LH, Total Testosterone levels were evaluated.
  Interventions: Procedure: TEP
- Lichtenstein repair: Lichtenstein method was performed to repair inguinal hernia . Patients were evaluated preoperatively, at 1 month and 6 months postoperatively, International Sexual Function Index (IFIF), International Prostatic Symptom Score, SF-36 Quality of Life Scale, Visual Analog Pain Scale, Beck Depression Scale, Inguinal Region Discrimination Test ( DT), DN4 Neuropathic Pain Survey, Uroflowmetry and FSH, LH, Total Testosterone levels were evaluated.
  Interventions: Procedure: Lichtenstein repair

INTERVENTIONS:
Procedure: TEP — By making a 2 cm incision under the umbilicus, skin subcutaneous tissues are passed through blunt dissections and the anterior fascia of the rectus muscle is exposed. An anterior rectus sheath with a scalpel is performed with a 15 mm incision. The rectus muscle is laterally lateralized and the balloon trocar or laparoscope itself is advanced from the midline to the symphysis pubis via the posterior rectus sheath. After the peritoneal cavity is dissected, a low pressure pneumoperitone 10 mm Hasson trocar or another 10 mm balloon caged trocar is advanced through the subumblic incision. 9-11 mmHg low pressure pneumoperitoneum is created to prevent the development of subcutaneous emphysema. For proper imaging, the patient should have complete muscle relaxation. The patient is given a position towards the light trandelenburg and non-hernia side.
  Groups: Total Extraperitoneal Repair
Procedure: Lichtenstein repair — After the inguinal incision, the skin and subcutaneous camper and scarpa tissues are passed and the external oblique aponeurosis is dissected in the direction of the extension of the fibers and the medial lateral edge of the rectus is dissected to the lateral inguinal ligament, then the spermatic cord is released and suspended.The spermatic cord is separated from the inguinal canal.
  In indirect hernias, the hernia sac is dissected from the spermatic cord and rejected into the abdomen by high ligation. In direct hernia, the hernia sac is pushed in and the transverse fascia is sutured with 2-3 separe stitches.
  Groups: Lichtenstein repair

SUMMARY:
The superiority of laparoscopic inguinal hernia surgery over open surgery has been shown in many high patient-numbered studies with early return to work, less pain and good cosmetic results. The aim of this study is to determine the differences between two different methods in terms of sexual, sensory, quality of life and urinary results.

DETAILED DESCRIPTION:
Between July 2017 and January 2018, 42 sexually active male patients were randomized with Laparoscopic Total Extraperitoneal (TEP) method and Lichtenstein (LCH) method and repair of inguinal hernia. Patients were evaluated preoperatively, at 1 month and 6 months postoperatively, International Sexual Function Index (IFIF), International Prostatic Symptom Score, SF-36 Quality of Life Scale, Visual Analog Pain Scale, Beck Depression Scale, Inguinal Region Discrimination Test ( DT), DN4 Neuropathic Pain Survey, Uroflowmetry and FSH, LH, Total Testosterone levels were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral inguinal hernia (diagnosed by physical examination or imaging)
* Sexual Active
* Male gender
* aged between 18 and 65
* ASA 1-2
* EHS Classification (Primary, lateral or medial, 1 and 2)

Exclusion Criteria:

* Patients with previous abdominal and inguinal hernia surgery
* ASA 3-4
* Sexually inactive
* Emergency patients (Etrangule inguinal hernia)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SEXUAL ACTIVE
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
International Sexual Function Index (IFIF) | UP TO 6 MONTHS
  Patients were evaluated preoperatively, at 1 month and 6 months postoperatively.Total 15 questions are included.Answers are include 1-5 options. (1:never , 5:always) Question 1,2,3,4,5,15 for erectile function , Question 9,10 for orgasm function , Question 11,12 for sexual desire , Question 6,7,8 for sexual satisfaction , Question 13,14 for general satisfaction.
International Prostatic Symptom Score | UP TO 6 MONTHS
  Patients were evaluated preoperatively, at 1 month and 6 months postoperatively. Total 7 questions which are about urinary functions are included.Answers are include 1-5 options. (1:never , 5:always) . Questions are :
  1. what is your frequency of feeling that your bladder does not empty after urination
  2. what is the frequency of needing to urinate in less than 2 hours after urination?
  3. what is your frequency of stopping several times when you urinate and restart?
  4. how often do you have difficulty urinating?
  5. how often did you feel the reduction in the power of your urine?
  6. how often have you experienced difficulty urinating?
  7. how many times have you gone to urinate until you get up in the morning?
SF-36 Quality of Life Scale | UP TO 6 MONTHS
  Patients were evaluated preoperatively, at 1 month and 6 months postoperatively
Visual Analog Pain Scale | UP TO 6 MONTHS
  Patients were evaluated preoperatively, at 1 month and 6 months postoperatively.pain scores (VAS: from 0 to 10, 0 = no pain, 10 = the worst pain) The higher score idicates the worse outcome.
Beck Depression Scale | UP TO 6 MONTHS
  Patients were evaluated preoperatively, at 1 month and 6 months postoperatively
Inguinal Region Discrimination Test ( DT) | UP TO 6 MONTHS
  Patients were evaluated preoperatively, at 1 month and 6 months postoperatively
DN4 Neuropathic Pain Survey | UP TO 6 MONTHS
  Patients were evaluated preoperatively, at 1 month and 6 months postoperatively. There are 4 questions in this survey and includes totally 10 points in it. Above the 4 points mean it is a neuropathic pain.
Uroflowmetry test for urination | UP TO 6 MONTHS
  In our study, the evaluation of urinary functions was performed with urolowmetry. Patients were evaluated preoperatively, at 1 month and 6 months postoperatively Voiding flow rates and voiding volumes were compared before and after surgery with Uroflowmetry
Follicle Stimulating Hormone levels | UP TO 6 MONTHS
  Patients were evaluated preoperatively, at 1 month and 6 months postoperatively
Luteinising Hormone levels | UP TO 6 MONTHS
  Patients were evaluated preoperatively, at 1 month and 6 months postoperatively
Total Testosterone levels | UP TO 6 MONTHS
  Patients were evaluated preoperatively, at 1 month and 6 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided